CLINICAL TRIAL: NCT04918030
Title: STaged Interventional Strategies for Acute ST-seGment Elevation Myocardial Infarction Patient With Multi-vessel Disease （STAGED）
Brief Title: STaged Interventional Strategies for Acute ST-seGment Elevation Myocardial Infarction Patient With Multi-vessel Disease（STAGED）
Acronym: SAGED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Collaborators: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yan Wang, Prof, Xiamen Cardiovascular Hospital, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020YLK14
Record Dates: First submitted 2021-05-24; First posted 2021-06-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: STEMI; Multi Vessel Coronary Artery Disease; Percutaneous Coronary Intervention; AMI Patients With Multivessel Disease, Staged PCI
Keywords: AMI, multivessel disease, PCI, staged complete revascularization
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early staged group (Active Comparator): Patients randomized to Early group will undergo staged PCI for all significant non-culprit lesions at 7±3 days after revascularization of the culprit lesion.
  Interventions: Procedure: Early staged PCI
- Late staged PCI (Experimental): Patients randomized to Late Group will undergo staged PCI for all significant non-culprit lesion at 30±15 days after primary PCI for culprit coronary lesions.
  Interventions: Procedure: Late staged PCI

INTERVENTIONS:
Procedure: Early staged PCI — After revascularization of the culprit lesion, all significant non-culprit vessel will be complete revascularzed during index the index procedure (7±3 day).
  Other Names: Percutaneous coronary intervention
  Arms: Early staged group
Procedure: Late staged PCI — During the index procedure, patients will have treated with primary PCI the culprit lesion only. Patients will be hospitalized again after 30±15 days to undergo PCI of the other significant coronary lesions.
  Other Names: Percutaneous coronary intervention
  Arms: Late staged PCI

SUMMARY:
An investigator-initiated, randomized, multicenter, two-arm, open-label study of consecutive patients presenting with STEMI and MVD Objectives: The present study aimed to investigate the difference in major adverse cardiac event (MACE) between Early staged PCI versus Late staged PCI groups among patients with ST-segment elevated myocardial infarction （STEMI and multi-vessel Disease（MVD) who underwent primary PCI using DES for culprit lesions.

Background: In patients with STEMI with MVD who underwent primary PCI, complete revascularization for non-culprit lesions has proved to reduce the risk of cardiovascular death and myocardial infarction. However, the ideal timing point for staged PCI for nonculprit lesions remains uncertain.

DETAILED DESCRIPTION:
A total of 1586 subjects with STEMI who met inclusion criteria and had no any exclusion criterion will be randomized (at a 1:1 ratio) to Early staged PCI group and Late staged PCI group. After successful percutaneous coronary intervention for culprit lesion, staged PCI for all non-culprit vessel with significant lesion defined at least 80% diameter stenosis by visual estimation and accompanied by a QFR measurement of less than or equal to 0.80 will be performed. Patients will be ranmized to the following groups at 1:1 ratio:

1. Patients randomized to the in-hospital staged PCI (Early group) will undergo PCI for all significant non-culprit lesions at 7±3 days after revascularization of the culprit lesion.
2. Patients randomized to out-hospital staged complete revascularization (Late group) will undergo PCI for all significant non-culprit lesions at 30±15 days after primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Established indication to PPCI according to the guidelines of American Heart Association and American College of Cardiology;
* Spontaneous acute STEMI (patients presenting within 24 hours of symptom onset) with MVD after successful revascularization of the culprit artery;
* De novo coronary lesion,
* TIMI Flow 3 ( Cases with TIMI flow 2 need to perform angiographic again in 24h ensured TIMI flow 3 for enrolling case )after revascularization of the culprit artery, residual stenosis ≤20% and no coronary dissection greater than or equal to type C leading to (threatening) vessel closure.
* At least one non-culprit coronary stenosis ≥ 80% and accompanied by QFR ≤0.8 in a vessel with a lumen diameter ≥2.5;

Exclusion Criteria:

* Age <18 yr and >80 yr;
* Cardiac shock, multiple organ failure, cerebral hemorrhage, severe aortic stenosis and myocardial infarction complications(cardiac rupture, ventricular septal rupture and papillary muscle rupture);
* Killip classification >3, cardiognic shock, shore-infarction of culprit artery after emergency PCI in 24 hours;
* Previous documented allergic reaction to drug and device of this study;
* Planned major surgery within 6 weeks in which impact DAPT;
* Participation in another clinical study, interfering with this protocol Uncertain;
* Life expectancy < 1 year;
* Any condition likely to interfere with study processes including follow-up visits or increase of risk accessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1586 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE), defined as cardiovascular death, MI, ischemia-driven revasculrization (for both culprit and non-culprit lesions). | 12 months
  The difference in MACE will be calculated from randomisation to 12 months.

SECONDARY OUTCOMES:
All-cause death | 12 months
  It will be calculated from randomisation to 12 months.
Myocardial Infarction (MI) | 12 months
  It will be calculated and compared from randomisation to 12 months Periprocedural MI (PMI): Defined as a CK-MB elevation greater than 10 times the upper reference limit (URL) within 72 hours post-procedure, in the absence of symptoms or ECG changes. If the patient presented with ischemic symptoms, ischemic ECG changes, or intra-procedural slow-flow or side-branch occlusion, PMI is defined as a CK-MB elevation greater than 5 times the URL.
  Spontaneous MI: Defined as a rise of cardiac biomarkers, preferably cardiac troponin (cTn), with at least one value above the 99th percentile URL, accompanied by at least one of the following: ischemic symptoms, new ischemic ECG changes (including new ST-T changes or new left bundle branch block), development of pathological Q waves, or imaging evidence of new regional wall motion abnormalities or loss of viable myocardium.
Revascularization | 12 months
  Ischemia-driven Coronary Revascularization Ischemia-driven coronary revascularization was defined in accordance with the Academic Research Consortium-2 (ARC-2) consensus. In this study, ischemia-driven coronary revascularization included any repeat percutaneous coronary intervention or coronary artery bypass grafting performed due to myocardial ischemia, irrespective of whether the lesion was located in a target or non-target vessel. Following the ARC-2 criteria, revascularization was considered ischemia-driven if it was associated with objective evidence of myocardial ischemia, including recurrent ischemic symptoms, ischemic changes on electrocardiogram, positive results from non-invasive stress testing, or fractional flow reserve less than or equal to 0.80. When functional assessment was not available, adjudication by the Clinical Events Committee using independent quantitative coronary angiography of baseline and repeat angiograms was required.
Cardiovascular death | 12 months
  Cardiovascular death includes sudden cardiac death, death due to acute myocardial infarction, heart failure, cerebrovascular events, other cardiovascular causes, such as pulmonary embolism, aortic disease, or complications arising from cardiovascular interventions or surgeries.
Heart failure-induced rehospitalization | 12 months
  Rate of New hospitalization for heart failure
Stroke | 12month
  According to the 2013 AHA/ASA guidelines, stroke is defined as cerebral infarction, intracerebral hemorrhage (ICH), or subarachnoid hemorrhage (SAH), all characterized by acute, focal dysfunction of the central nervous system (CNS) resulting from vascular causes.
Rate of contrast-induced nephropathy（CIN） | 12 months
  Contrast-Induced Nephropathy (Based on KDIGO criteria)
  1. An increase in serum creatinine to ≥1.5 times the baseline value within 7 days following exposure to contrast media.
  2. An absolute increase in serum creatinine of >0.3 mg/dL (26.5 μmol/L) within 48 hours after contrast exposure.
  3. Urine output <0.5 mL/kg/h for at least 6 consecutive hours post-procedure.

OTHER OUTCOMES:
Stent thrombosis | 12 months
  Stent Thrombosis (Based on Academic Research Consortium criteria)
  1. Definite ST: Clinical presentation of acute coronary syndrome with angiographic or pathological confirmation.
  2. Probable ST: Unexplained death within 30 days or acute ischemia in the target vessel territory without angiographic confirmation.
  3. Possible ST: Unexplained death after 30 days post-PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Dr, Principal Investigator — Clinical Trial Center of Xiamen Cardiovascular Hospital
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Data sharing could be considered upon the proposal was approved
Supporting Information: Analytic Code
Time Frame: One year lafter since publication
Access Criteria: All can access via reaching to PIs

REFERENCES:
- [Derived] Chen X, Li S, Wang B, Chen G, Yao Y, He Y, Wu X, Yang Y, Kang H, Ding L, Cheng Y, Shen Q, Guo H, Wang J, Wen S, Zhu L, Xing Y, Tong Q, Li P, Liu Y, Peng X, Chen SL, Wang Y. Staged interventional strategies for acute ST-segment elevation myocardial infarction patient with multi-vessel disease: Rationale and design of a multicenter, randomized STAGED trial. Am Heart J. 2026 Jan 13:107352. doi: 10.1016/j.ahj.2026.107352. Online ahead of print. PMID 41539383